CLINICAL TRIAL: NCT01599364
Title: Safety and Efficacy of Switching a Stable Combined Antiretroviral Therapeutic Regimen to Atazanavir With Ritonavir Plus Lamivudine in Treatment Experienced HIV Positive Patients With Full and Stable Virological Suppression
Brief Title: Atazanavir/r + Lamivudine Dual Therapy
Acronym: ATLAS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Simona Di Giambenedetto, MD, Catholic University of the Sacred Heart
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ATLAS 2; 2011-001060-21 (EudraCT Number)
Record Dates: First submitted 2012-05-14; First posted 2012-05-16 (Estimated); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Human Immunodeficiency Virus
Keywords: HIV infection; Atazanavir; Lamivudine; Ritonavir; virological suppression; non-inferiority; Combined antiretroviral therapy
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; HIV Infections | interventions — Atazanavir Sulfate; Ritonavir; Lamivudine; halofantrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Switch (Experimental): Switch to Atazanavir 300 mg with ritonavir 100 mg plus lamivudine 300 mg
  Interventions: Drug: Atazanavir, ritonavir, lamivudine
- continue (No Intervention): Continue Atazanavir 300 mg with ritonavir 100 mg with the same NRTI backbone

INTERVENTIONS:
Drug: Atazanavir, ritonavir, lamivudine — Lamivudine 300 mg 1 pill once-a-day, atazanavir 300 mg 1 pill with ritonavir 100 mg 1 pill once-a-day, taken together orally with a light meal
  Other Names: Lamivudine (Epivir, GSK), Atazanavir (Reyataz, BMS), Ritonavir (Norvir, Abbott)
  Arms: Switch

SUMMARY:
The purpose of this study is to evaluate the virological efficacy of maintenance therapy with atazanavir with ritonavir combined with lamivudine in treatment experienced HIV positive patients with full and stable virological suppression.

DETAILED DESCRIPTION:
The introduction of combined antiretroviral therapy (cART) dramatically improved the prognosis of HIV infection [1]; nowadays, virological suppression (viral load < 50 copies/mL) can be obtained in the vast majority of patients receiving cART. Nevertheless, antiretroviral drugs have short- and long-term side effects mainly regarding mitochondrial toxicity, impaired lipid and glucose metabolism, impairment of renal function and bone density and may contribute to increase the patients' cardiovascular risk.

Current treatment guidelines recommend three drug regimens with a "backbone" of 2 nucleos(t)ide reverse transcriptase inhibitors (N(t)RTIs) and a "third drug" to be chosen among non-nucleoside reverse transcriptase inhibitors (NNRTIs) and ritonavir-boosted protease inhibitors (PIr). Regimens containing less than three antiretroviral drugs are currently not recommended based on the high risk of virological failure and selection of drug resistance mutations (DRM) with previous experience of NRTI-only based approaches with the exception of boosted PIs monotherapy which is optional in patients with intolerance to NRTIs or requiring treatment simplification provided that they never experienced virological failures or admitted in exceptional circumstances.

Nevertheless, the investigation of possible new treatment paradigms remains attractive due to the high potency and low risk of selection of drug resistance mutations with PIr based therapies and the established long term toxicity of even newer and currently preferred N(t)RTIs, in particular the renal and bone toxicity of tenofovir and the debated potential association with increased cardiovascular risk of abacavir, which has been described in some cohort studies. Studies evaluating N(t)RTI-sparing treatment strategies are thus increasing in order to try to respond to the unmet medical needs of HIV-infected patients with metabolic complications and increasing risk of cardiovascular or renal diseases.

These studies will need to investigate the safety and efficacy of these alternative strategies, also evaluating their possible effects on renal function, bone mass density and risk of premature osteoporosis.

Atazanavir with ritonavir is a generally well tolerated lipid-friendly protease inhibitor with mild effects on lipid metabolism even when combined with low-dose ritonavir and is the only drug who achieved a non-significant difference in virological efficacy compared to efavirenz; like all other PIr-based regimens, failure of an atazanavir/ritonavir containing cART seems to protect against the development of drug resistance mutations to both the PI and the backbone. Lamivudine is a well tolerated NRTI which showed no significant toxicity in the short and long term and, together with its analog emtricitabine, is now a preferred option in most of the major international treatment guidelines; it has a good CNS penetration score and its only signature resistance mutation (M184V) deeply impairs the viral fitness and does not compromise the future treatment options.

The combination of these two drugs could therefore be an appealing possibility for treatment switch in stably virologically suppressed treatment-experienced patients with toxicity-related issues. The results of a previously planned 24 weeks interim analysis of a monocentric 48 weeks Italian pilot study evaluating this strategy in 40 patients has recently been presented at IAS conference in Vienna and showed no virologic failures without any "blip" and good tolerability with a significant improvement of renal function as measured by MDRD. These data look very promising and allow us to be confident in designing a randomized study in order to confirm these findings.

ELIGIBILITY:
Inclusion Criteria

* HIV positive patients 18 years of age or older who signed an informed consent form
* Already on cART, without any treatment interruption.
* Treated with a cART regimen containing atazanavir boosted with ritonavir since at least 3 months
* With full virological suppression (VL<50 copies/mL) for a minimum of six months and in at least in two consecutive determination 3 months +/-2 weeks apart from each other
* With CD4 cell count >200 since at least 6 months and without opportunistic infections or other AIDS-related events since at least one year before screening

Exclusion Criteria:

* Previous virological failure on a lamivudine- or PI-containing regimen or previous exposure to lamivudine-containing suboptimal antiretroviral regimens
* Patients with at least a single viral load blip over 200 copies/mL
* Patients with M184V or major atazanavir resistance mutation at previous genotypic resistance test (historical genotype)
* Pregnancy or lactation, planned pregnancy in the short-term
* Patients with HBsAg positive chronic HBV infection
* Patients who experienced major toxicities related to any of the study drugs in the past
* Patients with grade 4 laboratory abnormalities at baseline (excluding lipid profile and plasma bilirubin concentration).
* Patients with non-AIDS related illnesses which could, in the Clinician's judgement, jeopardize the patient's compliance to the study procedures (i.e. Child-Pugh B or higher liver cirrhosis, active cancers on treatment…).
* Patients treated with proton-pump inhibitors or other concomitant medication with potential for interactions reducing exposure to atazanavir

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 266 (Actual)
Dates: Start 2014-04; Primary Completion 2016-04 (Actual); Study Completion 2018-02-23 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with viral load < 50 copies/mL | at week 48
  Proportion of patients with viral load < 50 copies/mL at week 48 at the intention-to-treat with switch = failure analysis

SECONDARY OUTCOMES:
Efficacy and the safety of atazanavir with ritonavir combined with lamivudine in treatment experienced HIV positive patients with full and stable virological suppression | 48 and 96 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mauro MM Moroni, MD, Study Chair — Università di Milano Direttore clinica Malattie infettive; Pierluigi PZ Zoccolotti, MD, Study Chair — Università di Roma La Sapienza Dipartimento di Psicologia; Stafano SV Vella, MD, Study Chair — Dipartimento del farmaco all'Istituto Superiore della Sanità; Roberto RC Cauda, MD, Principal Investigator — Università Cattolica del S. Cuore Policlinico Universitario A. Gemelli
Locations (21):
- Italy (21):
  - Ospedale S. M. Annunziata - U.O. Malattie Infettive, Bagno a Ripoli, Firenze
  - P.O. "S. Caterina Novella" - UOC di Malattie Infettive, Galatina, Lecce
  - Azienda Ospedaliero Universitaria - Ospedali Riuniti di Ancona Struttura Organizzativa Dipartimentale (S.O.D) Clinica di Malattie infettive, Ancona
  - Azienda Ospedaliera Spedali Civili - Istituto di Malattie Infettive e Tropicali, Brescia
  - Azienda Ospedaliera di Rilievo Nazionale di alta specializzazione Garibaldi di Catania - Istituto Malattie infettive, Catania
  - Azienda Ospedaliera Universitaria San Martino - Clinica Malattie Infettive, Genova
  - A.O. Ospedale Niguarda Cà Granda - Malattie Infettive, Milan
  - Ospedale San Raffaele, Milan
  - Ospedale Luigi Sacco di Milano - Malattie infettive I Divisione, Milan
  - Ospedale Luigi Sacco di Milano Azienda ospedaliera e Polo Universitario - Dip. di Scienze Cliniche L. Sacco / Sez. Malattie Infettive, Milan
  - A.O. Universitaria Policlinico Paolo Giaccone di Palermo - Malattie Infettive, Palermo
  - Ospedale S. Maria della Misericordia, Perugia
  - IRCCS Istituto Dermatologico S. Gallicano (IFO) - UOC Dermatologia Infettiva, Roma
  - I.N.M.I. L. Spallanzani I.R.C.C.S. - .O.C. Malattie Infettive e Tropicali IV Divisione, Roma
  - I.N.M.I. L. Spallanzani I.R.C.C.S. - U.O.C. Infezioni Sistemiche e dell'Immunodepresso II Divisione, Roma
  - Università' degli studi di Roma La Sapienza - Dipartimento di Malattie Infettive e Tropicali, Roma
  - Università Cattolica del S. Cuore Policlinico Universitario A. Gemelli - Istituto di Clinica delle Malattie Infettive, Roma
  - Università degli studi di Sassari - Reparto Malattie Infettive, Sassari
  - Ospedale Amedeo di Savoia - Divisione A Malattie Infettive, Torino
  - Azienda ULSS 9 Treviso Ospedale S. Maria di Ca'Foncello - U.O. Malattie infettive, Treviso
  - Azienda Ospedaliera Universitaria Integrata di Verona - U.O.C. Malattie infettive, Verona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fabbiani M, Gagliardini R, Ciccarelli N, Quiros Roldan E, Latini A, d'Ettorre G, Antinori A, Castagna A, Orofino G, Francisci D, Chinello P, Madeddu G, Grima P, Rusconi S, Del Pin B, Lombardi F, D'Avino A, Foca E, Colafigli M, Cauda R, Di Giambenedetto S, De Luca A; ATLAS-M Study Group. Atazanavir/ritonavir with lamivudine as maintenance therapy in virologically suppressed HIV-infected patients: 96 week outcomes of a randomized trial. J Antimicrob Chemother. 2018 Jul 1;73(7):1955-1964. doi: 10.1093/jac/dky123. PMID 29668978
- [Derived] Di Giambenedetto S, Fabbiani M, Quiros Roldan E, Latini A, D'Ettorre G, Antinori A, Castagna A, Orofino G, Francisci D, Chinello P, Madeddu G, Grima P, Rusconi S, Di Pietro M, Mondi A, Ciccarelli N, Borghetti A, Foca E, Colafigli M, De Luca A, Cauda R; Atlas-M Study Group. Treatment simplification to atazanavir/ritonavir + lamivudine versus maintenance of atazanavir/ritonavir + two NRTIs in virologically suppressed HIV-1-infected patients: 48 week results from a randomized trial (ATLAS-M). J Antimicrob Chemother. 2017 Apr 1;72(4):1163-1171. doi: 10.1093/jac/dkw557. PMID 28093483
- See also: Related Info — http://atlas.cr-technology.com/